CLINICAL TRIAL: NCT06877182
Title: Novel Neuroradiological Workflow for the Assisted DIAgnosis and Management of DEMentia with Artificial Intelligence
Acronym: DIADEMA
Status: Active, not recruiting | Type: Observational
Sponsor: IRCCS SYNLAB SDN (Other)
Collaborators: UNINA (Unknown); UNITO (Unknown); Ospedale Fate bene Fratelli di Brescia (Unknown)
Responsible Party: Sponsor
Other Study IDs: 1/24
Record Dates: First submitted 2025-03-10; First posted 2025-03-14 (Actual); Last update posted 2025-03-19 (Actual); Status verified 2025-03

CONDITIONS: Alzheimer Disease; Dementia
Keywords: Neuroimaging; Artificial Intelligence (AI); Dementia; Assisted Diagnosis; Magnetic Resonance Imaging (MRI)
MeSH Terms: conditions — Alzheimer Disease; Dementia | interventions — Magnetic Resonance Imaging

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Diagnostic Test: Magnetic Resonance Imaging with Contrast — To evaluate the possibility to improve the neuroradiologic workflow with AI models

SUMMARY:
Identifying, screening and monitoring individuals at risk of Alzheimer's disease (AD) and dementia is a formidable challenge. Neuroimaging, and in particular magnetic resonance imaging (MRI), is crucial to detect structural neurodegeneration. However, current quantification tools are mainly limited to research contexts and produce non-standardised results. DIADEMA will build a systematic and standardised workflow to support neuro(radio)logical diagnosis. By combining artificial intelligence (AI) and machine learning (ML) the investigators will significantly enhance the clinical diagnosis of AD in neuroradiology. The investigator's main hypothesis is that an efficient workflow and associated higher diagnostic accuracy will substantially reduce healthcare costs, support clinical decision-making, provide second-opinion tools and improve patient care. This dual advance will have a profound impact on the healthcare system, marking an important step in the fight against Alzheimer's disease and dementia.

ELIGIBILITY:
Inclusion Criteria:

* patients who perform brain magnetic resonance during the last 20 years

Exclusion Criteria:

-

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients who perform brain magnetic resonance during the last 20 years
Sampling Method: Non-Probability Sample
Enrollment: 80000 (Estimated)
Dates: Start 2024-08-30 (Actual); Primary Completion 2025-12-30 (Estimated); Study Completion 2027-08-31 (Estimated)

PRIMARY OUTCOMES:
Improvement of the neuroradiological workflow performance | 1-36 month
  ROC curves

CONTACTS AND LOCATIONS:
Overall Officials: Marco Aiello, Principal Investigator — IRCCS SYNLAB SDN
Locations (1):
- Irccs Synlab Sdn, Naples, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Filip AC, Azevedo T, Passamonti L, Toschi N, Lio P. A novel Graph Attention Network Architecture for modeling multimodal brain connectivity. Annu Int Conf IEEE Eng Med Biol Soc. 2020 Jul;2020:1071-1074. doi: 10.1109/EMBC44109.2020.9176613. PMID 33018171
- [Background] Spasov SE, Passamonti L, Duggento A, Lio P, Toschi N. A Multi-modal Convolutional Neural Network Framework for the Prediction of Alzheimer's Disease. Annu Int Conf IEEE Eng Med Biol Soc. 2018 Jul;2018:1271-1274. doi: 10.1109/EMBC.2018.8512468. PMID 30440622
- [Background] Spasov S, Passamonti L, Duggento A, Lio P, Toschi N; Alzheimer's Disease Neuroimaging Initiative. A parameter-efficient deep learning approach to predict conversion from mild cognitive impairment to Alzheimer's disease. Neuroimage. 2019 Apr 1;189:276-287. doi: 10.1016/j.neuroimage.2019.01.031. Epub 2019 Jan 14. PMID 30654174
- [Background] Esteban O, Birman D, Schaer M, Koyejo OO, Poldrack RA, Gorgolewski KJ. MRIQC: Advancing the automatic prediction of image quality in MRI from unseen sites. PLoS One. 2017 Sep 25;12(9):e0184661. doi: 10.1371/journal.pone.0184661. eCollection 2017. PMID 28945803
- [Background] van Leeuwen KG, Schalekamp S, Rutten MJCM, van Ginneken B, de Rooij M. Artificial intelligence in radiology: 100 commercially available products and their scientific evidence. Eur Radiol. 2021 Jun;31(6):3797-3804. doi: 10.1007/s00330-021-07892-z. Epub 2021 Apr 15. PMID 33856519
- [Background] Archetti D, Young AL, Oxtoby NP, Ferreira D, Martensson G, Westman E, Alexander DC, Frisoni GB, Redolfi A; for Alzheimer's Disease Neuroimaging Initiative and EuroPOND Consortium. Inter-Cohort Validation of SuStaIn Model for Alzheimer's Disease. Front Big Data. 2021 May 20;4:661110. doi: 10.3389/fdata.2021.661110. eCollection 2021. PMID 34095821
- [Background] Redolfi A, De Francesco S, Palesi F, Galluzzi S, Muscio C, Castellazzi G, Tiraboschi P, Savini G, Nigri A, Bottini G, Bruzzone MG, Ramusino MC, Ferraro S, Gandini Wheeler-Kingshott CAM, Tagliavini F, Frisoni GB, Ryvlin P, Demonet JF, Kherif F, Cappa SF, D'Angelo E. Medical Informatics Platform (MIP): A Pilot Study Across Clinical Italian Cohorts. Front Neurol. 2020 Sep 23;11:1021. doi: 10.3389/fneur.2020.01021. eCollection 2020. PMID 33071930
- [Background] Ribaldi F, Altomare D, Jovicich J, Ferrari C, Picco A, Pizzini FB, Soricelli A, Mega A, Ferretti A, Drevelegas A, Bosch B, Muller BW, Marra C, Cavaliere C, Bartres-Faz D, Nobili F, Alessandrini F, Barkhof F, Gros-Dagnac H, Ranjeva JP, Wiltfang J, Kuijer J, Sein J, Hoffmann KT, Roccatagliata L, Parnetti L, Tsolaki M, Constantinidis M, Aiello M, Salvatore M, Montalti M, Caulo M, Didic M, Bargallo N, Blin O, Rossini PM, Schonknecht P, Floridi P, Payoux P, Visser PJ, Bordet R, Lopes R, Tarducci R, Bombois S, Hensch T, Fiedler U, Richardson JC, Frisoni GB, Marizzoni M. Accuracy and reproducibility of automated white matter hyperintensities segmentation with lesion segmentation tool: A European multi-site 3T study. Magn Reson Imaging. 2021 Feb;76:108-115. doi: 10.1016/j.mri.2020.11.008. Epub 2020 Nov 19. PMID 33220450
- [Background] Morid MA, Borjali A, Del Fiol G. A scoping review of transfer learning research on medical image analysis using ImageNet. Comput Biol Med. 2021 Jan;128:104115. doi: 10.1016/j.compbiomed.2020.104115. Epub 2020 Nov 13. PMID 33227578
- [Background] Bao S, Boyd BD, Kanakaraj P, Ramadass K, Meyer FAC, Liu Y, Duett WE, Huo Y, Lyu I, Zald DH, Smith SA, Rogers BP, Landman BA. Integrating the BIDS Neuroimaging Data Format and Workflow Optimization for Large-Scale Medical Image Analysis. J Digit Imaging. 2022 Dec;35(6):1576-1589. doi: 10.1007/s10278-022-00679-8. Epub 2022 Aug 3. PMID 35922700
- [Background] Rajput D, Wang WJ, Chen CC. Evaluation of a decided sample size in machine learning applications. BMC Bioinformatics. 2023 Feb 14;24(1):48. doi: 10.1186/s12859-023-05156-9. PMID 36788550
- [Background] McKhann GM, Knopman DS, Chertkow H, Hyman BT, Jack CR Jr, Kawas CH, Klunk WE, Koroshetz WJ, Manly JJ, Mayeux R, Mohs RC, Morris JC, Rossor MN, Scheltens P, Carrillo MC, Thies B, Weintraub S, Phelps CH. The diagnosis of dementia due to Alzheimer's disease: recommendations from the National Institute on Aging-Alzheimer's Association workgroups on diagnostic guidelines for Alzheimer's disease. Alzheimers Dement. 2011 May;7(3):263-9. doi: 10.1016/j.jalz.2011.03.005. Epub 2011 Apr 21. PMID 21514250
- [Background] Boccardi M, Altomare D, Ferrari C, Festari C, Guerra UP, Paghera B, Pizzocaro C, Lussignoli G, Geroldi C, Zanetti O, Cotelli MS, Turla M, Borroni B, Rozzini L, Mirabile D, Defanti C, Gennuso M, Prelle A, Gentile S, Morandi A, Vollaro S, Volta GD, Bianchetti A, Conti MZ, Cappuccio M, Carbone P, Bellandi D, Abruzzi L, Bettoni L, Villani D, Raimondi MC, Lanari A, Ciccone A, Facchi E, Di Fazio I, Rozzini R, Boffelli S, Manzoni L, Salvi GP, Cavaliere S, Belotti G, Avanzi S, Pasqualetti P, Muscio C, Padovani A, Frisoni GB; Incremental Diagnostic Value of Amyloid PET With [18F]-Florbetapir (INDIA-FBP) Working Group. Assessment of the Incremental Diagnostic Value of Florbetapir F 18 Imaging in Patients With Cognitive Impairment: The Incremental Diagnostic Value of Amyloid PET With [18F]-Florbetapir (INDIA-FBP) Study. JAMA Neurol. 2016 Dec 1;73(12):1417-1424. doi: 10.1001/jamaneurol.2016.3751. PMID 27802513
- [Background] Jack CR Jr, Bennett DA, Blennow K, Carrillo MC, Feldman HH, Frisoni GB, Hampel H, Jagust WJ, Johnson KA, Knopman DS, Petersen RC, Scheltens P, Sperling RA, Dubois B. A/T/N: An unbiased descriptive classification scheme for Alzheimer disease biomarkers. Neurology. 2016 Aug 2;87(5):539-47. doi: 10.1212/WNL.0000000000002923. Epub 2016 Jul 1. PMID 27371494
- [Background] Teipel S, Grothe MJ; Alzheimer's Disease Neuroimaging Initiative. MRI-based basal forebrain atrophy and volumetric signatures associated with limbic TDP-43 compared to Alzheimer's disease pathology. Neurobiol Dis. 2023 May;180:106070. doi: 10.1016/j.nbd.2023.106070. Epub 2023 Mar 8. PMID 36898615
- [Background] De Francesco S, Galluzzi S, Vanacore N, Festari C, Rossini PM, Cappa SF, Frisoni GB, Redolfi A. Norms for Automatic Estimation of Hippocampal Atrophy and a Step Forward for Applicability to the Italian Population. Front Neurosci. 2021 Jun 28;15:656808. doi: 10.3389/fnins.2021.656808. eCollection 2021. PMID 34262425
- [Background] Hosny A, Parmar C, Quackenbush J, Schwartz LH, Aerts HJWL. Artificial intelligence in radiology. Nat Rev Cancer. 2018 Aug;18(8):500-510. doi: 10.1038/s41568-018-0016-5. PMID 29777175
- [Background] Qiu S, Miller MI, Joshi PS, Lee JC, Xue C, Ni Y, Wang Y, De Anda-Duran I, Hwang PH, Cramer JA, Dwyer BC, Hao H, Kaku MC, Kedar S, Lee PH, Mian AZ, Murman DL, O'Shea S, Paul AB, Saint-Hilaire MH, Alton Sartor E, Saxena AR, Shih LC, Small JE, Smith MJ, Swaminathan A, Takahashi CE, Taraschenko O, You H, Yuan J, Zhou Y, Zhu S, Alosco ML, Mez J, Stein TD, Poston KL, Au R, Kolachalama VB. Multimodal deep learning for Alzheimer's disease dementia assessment. Nat Commun. 2022 Jun 20;13(1):3404. doi: 10.1038/s41467-022-31037-5. PMID 35725739
- [Background] Faggioni L, Coppola F, Ferrari R, Neri E, Regge D. Usage of structured reporting in radiological practice: results from an Italian online survey. Eur Radiol. 2017 May;27(5):1934-1943. doi: 10.1007/s00330-016-4553-6. Epub 2016 Aug 29. PMID 27572812
- [Background] Bosco P, Redolfi A, Bocchetta M, Ferrari C, Mega A, Galluzzi S, Austin M, Chincarini A, Collins DL, Duchesne S, Marechal B, Roche A, Sensi F, Wolz R, Alegret M, Assal F, Balasa M, Bastin C, Bougea A, Emek-Savas DD, Engelborghs S, Grimmer T, Grosu G, Kramberger MG, Lawlor B, Mandic Stojmenovic G, Marinescu M, Mecocci P, Molinuevo JL, Morais R, Niemantsverdriet E, Nobili F, Ntovas K, O'Dwyer S, Paraskevas GP, Pelini L, Picco A, Salmon E, Santana I, Sotolongo-Grau O, Spiru L, Stefanova E, Popovic KS, Tsolaki M, Yener GG, Zekry D, Frisoni GB. The impact of automated hippocampal volumetry on diagnostic confidence in patients with suspected Alzheimer's disease: A European Alzheimer's Disease Consortium study. Alzheimers Dement. 2017 Sep;13(9):1013-1023. doi: 10.1016/j.jalz.2017.01.019. Epub 2017 Mar 3. PMID 28263741
- [Background] Buchlak QD, Milne MR, Seah J, Johnson A, Samarasinghe G, Hachey B, Esmaili N, Tran A, Leveque JC, Farrokhi F, Goldschlager T, Edelstein S, Brotchie P. Charting the potential of brain computed tomography deep learning systems. J Clin Neurosci. 2022 May;99:217-223. doi: 10.1016/j.jocn.2022.03.014. Epub 2022 Mar 12. PMID 35290937
- [Background] Redolfi A, Archetti D, De Francesco S, Crema C, Tagliavini F, Lodi R, Ghidoni R, Gandini Wheeler-Kingshott CAM, Alexander DC, D'Angelo E. Italian, European, and international neuroinformatics efforts: An overview. Eur J Neurosci. 2023 Jun;57(12):2017-2039. doi: 10.1111/ejn.15854. Epub 2022 Dec 14. PMID 36310103
- [Background] Kwee TC, Kwee RM. Workload of diagnostic radiologists in the foreseeable future based on recent scientific advances: growth expectations and role of artificial intelligence. Insights Imaging. 2021 Jun 29;12(1):88. doi: 10.1186/s13244-021-01031-4. PMID 34185175
- [Background] Aiello M, Cavaliere C, D'Albore A, Salvatore M. The Challenges of Diagnostic Imaging in the Era of Big Data. J Clin Med. 2019 Mar 6;8(3):316. doi: 10.3390/jcm8030316. PMID 30845692
- [Background] Aiello M, Esposito G, Pagliari G, Borrelli P, Brancato V, Salvatore M. How does DICOM support big data management? Investigating its use in medical imaging community. Insights Imaging. 2021 Nov 8;12(1):164. doi: 10.1186/s13244-021-01081-8. PMID 34748101
- [Background] Jonsson L, Tate A, Frisell O, Wimo A. The Costs of Dementia in Europe: An Updated Review and Meta-analysis. Pharmacoeconomics. 2023 Jan;41(1):59-75. doi: 10.1007/s40273-022-01212-z. Epub 2022 Nov 15. PMID 36376775